CLINICAL TRIAL: NCT06145815
Title: Predictive Model for Minimal Important Change After Rotator Cuff Repair Using Machine Learning Methods: A Pilot Study
Brief Title: Machine Learning Predictive Model for Rotator Cuff Repair Failure
Status: Completed | Type: Observational
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Orthopaedic Surgeon, La Tour Hospital
Other Study IDs: CCER #2020-02670
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rotator Cuff Tears
Keywords: Artificial intelligence; Machine Learning; Minimal Important Change
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIC RCR patients: Patients who improved their SANE score beyond the minimal important change one year after arthroscopic rotator cuff repair
  Interventions: Procedure: Arthroscopic rotator cuff repair
- No-MIC RCR patients: Patients who did not improve their SANE score beyond the minimal important change one year after arthroscopic rotator cuff repair
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — Patients underwent an arthroscopic repair for rotator cuff lesions

SUMMARY:
There is little overall evidence behind clinical practice guidelines for diagnosis and treatment of rotator cuff repair. The purpose of this study was to compare the performance of different machine learning models that use pre-operative data from an international and multicentric database to predict if a patient that underwent rotator cuff repair could achieve the minimal important change (MIC) for single assessment numeric evaluation (SANE) at one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primarily treated for rotator cuff tears by partial or complete surgical repair with a planned arthroscopic procedure
* Reparable tears
* No language barrier hindering questionnaire completion or legal incompetence were not included

Exclusion Criteria:

* missing pre- or post-operative single-assessment numeric evaluation (SANE)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who were primarily treated for rotator cuff tears by partial or complete surgical repair with a planned arthroscopic procedure were included in study.
Sampling Method: Non-Probability Sample
Enrollment: 4789 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
SANE score | At 12 post-operative months
  Single Assessment Numeric Evaluation (SANE). From 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour hospital, Meyrin (1217) Geneva, Switzerland
Locations (1):
- La Tour hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided